CLINICAL TRIAL: NCT04766866
Title: Protocol of the PE37 Study: A Multicenter Randomized Trial of Screening With sFlt1/PlGF and Planned Delivery to Prevent Preeclampsia at Term
Brief Title: sFlt1/PlGF and Planned Delivery to Prevent Preeclampsia at Term.
Acronym: PE37
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Elisa Llurba, Professor of Obstetric and Gynecology Universitat Autònoma de Barcelona, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PE37
Record Dates: First submitted 2021-02-08; First posted 2021-02-23 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Preeclampsia; Intrauterine Growth Restriction; Maternal Hypertension; Neonatal Outcome; Perinatal Death
Keywords: Preeclampsia, angiogenic factors, perinatal death, induction of labour
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation; Hypertension, Pregnancy-Induced; Perinatal Death | interventions — Pregnancy

STUDY DESIGN:
Intervention Model Description: Prospective, open-label randomized study with parallel groups.
Who Masked: Participant, Care Provider
Masking Description: Upon agreement to participate in this study, patients will be randomized to one of the following groups:
  • Intervention group or reveal group (sFlt-1/PlGF result known to clinicians). A ratio cutoff of >p90th will be used to define low and elevated risk of developing a placental complications of pregnancy and therefore induction of labour will be offered from 37th weeks of gestation Non-intervention or non-reveal (result unknown) group: routine follow-up and spontaneous delivery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-intervention or non-reveal group (No Intervention): Non-intervention or non-reveal (result unknown) group: routine follow-up and spontaneous delivery
- Intervention group or reveal group (Experimental): A ratio cutoff of >p90th will be used to define low and elevated risk of developing a placental complications of pregnancy and therefore induction of labour will be offered from 37th weeks of gestation
  Interventions: Diagnostic Test: sFlt1/PlGF screening in maternal blood at 35 to 36.6 weeks of gestation

INTERVENTIONS:
Diagnostic Test: sFlt1/PlGF screening in maternal blood at 35 to 36.6 weeks of gestation — A ratio cutoff of >p90th will be used to define low and elevated risk of developing a placental complications of pregnancy and therefore induction of labour will be offered from 37th weeks of gestation
  Arms: Intervention group or reveal group

SUMMARY:
* Preeclampsia (PE) affects ~5% of pregnancies. Although improved obstetrical care has significantly diminished associated maternal mortality, PE remains a leading cause of maternal morbidity and mortality in the world.
* Term PE accounts for 70% of all PE and a large proportion of maternal-fetal morbidity related with this condition. Prediction and prevention of term PE remains unsolved.
* Previously proposed approaches are based on combined screening and/or prophylactic drugs, but these policies are unlikely to be implementable in many world settings.
* Recent evidence shows that sFlt1-PlGF ratio at 35-37w predicts term PE with 80% detection rate.
* Likewise, recent studies demonstrate that induction of labor (IOL) from 37w is safe.
* The investigators hypothesize that a single-step universal screening for term PE based on sFlt1/PlGF ratio at 35-37w followed by IOL from 37w would reduce the prevalence of term PE without increasing cesarean section rates or adverse neonatal outcomes.
* The investigators propose a randomized clinical trial to evaluate the impact of a screening of term PE with sFlt-1/PlGF ratio in asymptomatic nulliparous women at 35-37w. Women will be assigned to revealed (sFlt-1/PlGF known to clinicians) versus concealed (unknown) arms. A cutoff of >90th centile will be used to define high risk of PE and offer IOL from 37w.
* If successful, the results of this trial will provide evidence to support a simple universal screening strategy reducing the prevalence of term PE, which could be applicable in most healthcare settings and have enormous implications on perinatal outcomes and public health policies worldwide.

DETAILED DESCRIPTION:
Finding an effective prediction and prevention for term PE remains an unsolved challenge. From previous recent evidence it seems clear that prediction very close to term may achieve a high detection rate, but there is no evidence as to which strategy might be effective in preventing PE in high-risk women. The investigators postulate that a solution that would be applicable in most settings worldwide would require a simplified, pragmatic, approach. The rationale of this proposal is that PE could be reduced with a single-step lab test screening followed by induction of labor (IOL).

A single-step lab measure to detect PE. Combined algorithms using angiogenic factors with Doppler ultrasound and maternal features seem to achieve the highest performance in detecting pre-clinical PE. However, the need to train staff and change pregnancy care protocols renders difficult generalization in high-resource and even more low-resource settings. On the contrary, single lab tests can be more easily incorporated into the mainstream clinical practice and provide a widespread solution for high-resource settings and specially sub-optimal healthcare systems heavily affected by the consequences of term PE. Angiogenic factors are the obvious candidate for these purposes. The sFlt1/PlGF ratio at 35-36w predicts term PE with a DR of 82% and is a standardized lab test nowadays, realizable by ELISA with widely available automated lab platforms. Normal values in late pregnancy have been reported and are fairly similar among different populations. As preliminary research for this study, the investigators have confirmed that the gestational-age adjusted normal values of sFlt1/PlGF matched quite remarkably those previously published in different populations across Europe. A one-step screening with sFlt1/PlGF would select a 5-10% of the population with the highest risk for PE.

IOL at 37 weeks as an intervention in women at high-risk for PE. Previous trials based on statins have failed to show a reduction of PE in high-risk women. IOL at 37 weeks is an alternative to avoid PE in those high-risk women. IOL has consistently been demonstrated to be safe ( ) and does not affect long-term maternal quality of life ( ). Both the HYPITAT and the DIGITAT randomized trials showed that IOL did not increase caesarean rates or adverse neonatal outcomes ( ). A recent large randomized trial in the US has shown that even in low-risk women, universal IOL decreased cesarean section rates and was well accepted ( ). While in low-risk pregnancies labour induction has been found to be beneficial from 39 weeks (ARRIVE study), in women with placental-related conditions such as hypertension (HYPITAT) or small-for-gestational age (DIGITAT) it is 37+ weeks when the trade-off between neonatal and maternal benefits makes induction recommendable.

Therefore, the investigators hypothesize that a single-step universal screening for term PE based on sFlt1/PlGF ratio at 35-36.6 w followed by IOL at 37w in those women found to be at high risk might represent a feasible and reproducible strategy, applicable worldwide, to reduce the prevalence of term PE without increasing cesarean section rates or adverse neonatal outcomes.

Individual participant data, study protocol, statistical analysis plan and informed consent form will be available with publication by email addresses after approval of a proposal with a signed data access agreement

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Singleton pregnancies
* >18 years old
* 35.0-36.6 weeks of gestation
* Maternal written consent form

Exclusion Criteria:

* Fetuses/neonates with major malformations or genetic anomalies that could modify the timing of delivery or has an impact on obstetric outcome
* Suspected fetal growth restriction (estimated fetal weight <3 centile or between the 3rd and 10th centile together with abnormal Doppler in the mean uterine artery Doppler pulsatility index, or in umbilical artery pulsatility index or in the middle cerebral artery or in the cerebral umbilical index (CPR))
* Participation in another interventional study that could modify the timing of delivery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 9132 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of term Preeclampsia development | 4 weeks
  Number of participants with term preeclampsia/total number participants.

SECONDARY OUTCOMES:
Maternal morbidity rate | 6 weeks
  Composite including any of the following: (i) HELLP syndrome; (ii) Central nervous system dysfunction (eclampsia, Glasgow Coma Score <13, stroke, reversible ischemic neurological deficit or cortical blindness); (iii) hepatic dysfunction; (iv) renal dysfunction; (v) respiratory dysfunction; (vi) cardiovascular dysfunction; (vii) placental abruption; or, (viii) a requirement for transfusion of blood products according to the total deliveries.
Maternal Hospital stay | 6 weeks
  Days of admission
Caesarean section rate | 4 weeks
  number of c-section / total deliveries
Perinatal complications rate | 18 weeks
  Presence of placental abruptio, severe fetal growth restriction (defined as birth weight <3rd centile), perinatal mortality, an Apgar score at 5-minute below 7.0, an umbilical artery pH below 7.10, need for respiratory support within 72 hours after birth neonatal intraventricular haemorrhage grade III/IV, necrotizing enterocolitis, sepsis, or hypoxic ischemic encephalopathy/total deliveries.
Neonatal hospital stay | 18 weeks
  Days
Maternal experience | 12 weeks
  Satisfaction score (PSS, STAI, WHO and Labor Agentry scale).
Incurred costs | 6 weeks
  Calculated costs
Number of participants with Cardiovascular risk | 6 months post-delivery
  Maternal blood pressure and endothelial function 6-months postpartum/ participants

CONTACTS AND LOCATIONS:
Locations (21):
- CHU Liège, Liège, Belgium
- Clinica del Prado SAS, Bogotá, Colombia
- Institute for the Care of Mother and Child, Prague, Czechia
- Medicina Fetal Quito, Quito, Ecuador
- India (3):
  - Maulana Azad Medical College (MAMC), New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences (AIIMS) Ansari Nagar, New Delhi, National Capital Territory of Delhi
  - Vardhman Mahavir Medical College (VMMC), New Delhi, National Capital Territory of Delhi
- Hospital Gineco-Obstetricia nº4, Mexico City, Mexico
- Hospital Santo Tomas, Panama City, Panama
- Centre of Postgraduate Medical Education, Obstetrics and Gynecology and Perinatal Medicine, Warsaw, Poland
- Spain (11):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas de Gran Canaria, Canary Islands
  - Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Maternitat del Clínic, Barcelona
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital La Paz, Madrid
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital la Fe, Valencia
  - Hospital Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Llurba E, Crispi F, Crovetto F, Youssef L, Delgado JL, Puig I, Mora J, Krofta L, Mackova K, Martinez-Varea A, Tubau A, Ruiz A, Paya A, Prat M, Chantraine F, Comas C, Kajdy A, Lopez-Tinajero MF, Figueras F, Gratacos E; PE37 study group. Multicentre randomised trial of screening with sFlt1/PlGF and planned delivery to prevent pre-eclampsia at term: protocol of the PE37 study. BMJ Open. 2024 Mar 8;14(3):e076201. doi: 10.1136/bmjopen-2023-076201. PMID 38458783